CLINICAL TRIAL: NCT04141124
Title: Effects of Relaxing Breathing Combined With Biofeedback on the Performance and Stress of Residents During a High-fidelity Simulation Session.
Brief Title: Effects of Relaxing Breathing Combined With Biofeedback on the Performance and Stress of Residents During HFS
Acronym: RETROSIMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, principal investigator, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RETROSIMU
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Stress, Psychological; Stress, Physiological; Performance Anxiety; Critical Incident
Keywords: medical education; simulated critical situation; stress management and performance
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: 3 paralel arms of interventions
Who Masked: Investigator, Outcomes Assessor
Masking Description: Intervention will not be observed by outcomes assessor Performance will be evaluated on video recording after the simulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): 5 minutes of reading fictitious biological medical results that are almost normal and unrelated to the upcoming scenario. This condition reflects a likely activity in relation to other patients in charge, pending an announced critical situation.
  Interventions: Other: Control
- Relaxing Breathing (Active Comparator): 5 minutes of relaxing breathing guided by a computer helping to follow inspiration and expiration.
  Interventions: Other: Relaxing Breathing
- Breathing exercise combined with HRV (Experimental): 5 minutes of relaxing breathing, guided by a computer helping to follow inspiration and expiration and coupled with direct biological feedback on HRV.
  Interventions: Other: breathing exercise/HRV-biofeedback

INTERVENTIONS:
Other: breathing exercise/HRV-biofeedback — 5 min of relaxing breathing, coupled with biological feedback.
  Other Names: 0
  Arms: Breathing exercise combined with HRV
Other: Relaxing Breathing — 5 minutes of relaxing breathing guided by a computer helping to follow inspiration and expiration.
  Arms: Relaxing Breathing
Other: Control — 5 minutes of reading fictitious biological medical results
  Arms: Control

SUMMARY:
The harmful effects of stress on health professionals are expressed both in terms of their health (physical or mental) and the quality of work (reduced memory capacity, deterioration in patient care). These adverse effects highlight the importance of implementing effective coping strategies and/or early learning of stress management methods in medical training programs.

Relaxation breathing techniques coupled with heart rate variability (HRV) biofeedback is one of the new techniques used to reduce the stress level.

No research has yet tested the effects of HRV induced by relaxation breathing technique before managing a simulated critical situation.

DETAILED DESCRIPTION:
This is a randomized, controlled study conducted at the university simulation centre in healthcare of Lyon, France. The high-fidelity simulation (HFS) will be used as a research tool and the topics included will be the HFS residents summoned to critical care situations as part of their training curriculum. The study has received prior approval from the UCBL1. Ethics Committee. After information (protocol and objective of the study), signature of consent, and one minute of relaxing breathing training, the residents as active participants in HFS, will be included in the study. They will be equipped with Hexoskin® jackets collecting heart rate, heart rate variability, breathing rate continuously and an Empathica® connected watch for continuous measurement of electrodermal activity. Then each resident will be randomized into one of the three intervention groups that are:

* a relaxing breathing exercise coupled with biofeedback
* a breathing exercise without biofeedback
* a control occupation (observation of normal biological results). Each intervention will last five minutes and will be conducted between the briefing and the scenario.

Main objective :

The objective of this study is to compare during HFS, the performance of residents during critical care scenarios. The performance analysis will be performed by two independent and blinded evaluators, based on the video recordings of scenarios. The overall performance will be the addition of technical skills (specific rating grid for each scenario on 100 pts) and non-technical skills assessed by the OTTAWA GRS grid (adjusted to 100 pts).

Secondary objectives :

* Compare the effects of the three interventions on reducing psychological stress.
* Compare the effects of the three interventions on reducing physiological stress.
* Compare the effects of the three interventions on increasing cardiac coherence scores.

ELIGIBILITY:
Inclusion Criteria:

* Adult person
* Registered in specialized diploma of medical training.
* Invited for a high-fidelity simulation session at the Lyon university simulation center.
* Have signed an informed consent form.

Exclusion Criteria:

* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Performance during HFS | day 0: during the HFS
  Technical specific performance for each scenario. Non-technical performance (with Ottawa GRS Grid).

SECONDARY OUTCOMES:
Physiological stress | day 0: during the HFS
  HRV
Psychological stress | 0: during the HFS
  Visual analog scales from 0 to 100 mm the higher the higher stress level
Individual psychological characteristics | 0: during the HFS
  Personality traits (Big-5)
psychological stress consequences | 0: during the HFS
  Activation-Desactivation Adjective Check List: for the four subscales: Energy, Tiredness, Tension , and Calmness
Individual psychological characteristics | 0: during the HFS
  Depressive symptoms (Beck) the higher the more depressive symptoms Anxiety-Trait (STAI-T)
Individual psychological characteristics | 0: during the HFS
  Fear of negative evaluation (PEN). from 0 to 30 the higher the more fear
Physiological stress | day 0: during the HFS
  electrodermal activity

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lilot, M.D., Principal Investigator — University of Lyon medical center Rockfeller
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schlatter ST, Therond CC, Guillot A, Louisy SP, Duclos A, Lehot JJ, Rimmele T, Debarnot US, Lilot ME. Effects of relaxing breathing paired with cardiac biofeedback on performance and relaxation during critical simulated situations: a prospective randomized controlled trial. BMC Med Educ. 2022 Jun 2;22(1):422. doi: 10.1186/s12909-022-03420-9. PMID 35655176